CLINICAL TRIAL: NCT02184442
Title: The PARTNER II Trial "Placement of AoRTic TraNscathetER" Valves Trial" (US) [PII B] for Inoperable Patients
Brief Title: The PARTNER II Trial: Placement of AoRTic TraNscathetER Valves - PII B
Acronym: PARTNERII B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Collaborators: American College of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-12-PIIB
Record Dates: First submitted 2014-01-17; First posted 2014-07-09 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Severe; Symptomatic; Calcific Aortic Stenosis
Keywords: SAPIEN; TAVR; THV; Aortic Stenosis; Heart Valve Disease; Aortic Valve; Retroflex; SAPIEN XT
MeSH Terms: conditions — Lymphoma, Follicular; Aortic Valve, Calcification of; Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TAVR - SAPIEN XT (Experimental): TAVR (transaortic valve replacement) with SAPIEN XT
  Interventions: Device: TAVR Implantation with SAPIEN XT
- TAVR - SAPIEN (Active Comparator): TAVR (transaortic valve replacement) with SAPIEN is the control arm
  Interventions: Device: TAVR Implantation with SAPIEN

INTERVENTIONS:
Device: TAVR Implantation with SAPIEN XT — Inoperable operable patients requiring the transcatheter aortic heart valve replacement
  Arms: TAVR - SAPIEN XT
Device: TAVR Implantation with SAPIEN — Inoperable operable patients requiring the transcatheter aortic heart valve replacement
  Arms: TAVR - SAPIEN

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the SAPIEN XT™ THV with the associated delivery system for inoperable patients with severe symptomatic native aortic stenosis.

DETAILED DESCRIPTION:
Cohort B was a 1:1 randomized, controlled study independently powered to compare transcatheter heart valve therapy with the first generation (SAPIEN™ THV) system to transcatheter heart valve therapy with the second generation (SAPIEN XT THV) system in patients who could not undergo surgery (inoperable).

Patients in the control arm of Cohort B received an Edwards SAPIEN THV with the associated delivery system while patients in the treatment arm of Cohort B received an Edwards SAPIEN XT THV with the associated delivery system.

ELIGIBILITY:
Inclusion Criteria

1. Patient was symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater.
2. The probability of death or serious, irreversible morbidity is greater than or equal to 50%.
3. The heart team agreed (and verified in the case review process) that valve implantation would likely benefit the patient.
4. The study patient or the study patient's legal representative was informed of the nature of the study, agreed to its provisions and had provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
5. The study patient agreed to comply with all required post-procedure follow-up visits including annual visits through 5 years and analysis close date visits, which was conducted as a phone follow-up.

Exclusion Criteria

1. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified.
2. Significant aortic disease, including marked tortuosity (hyperacute bend), aortic arch atheroma [especially if thick (> 5 mm), protruding or ulcerated] or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta. (Transfemoral)
3. Currently participating in an investigational drug or another device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
4. It is known that the patient is currently enrolled in the PARTNER I Trial or was withdrawn from the PARTNER I Trial prior to endpoint analysis.
5. Active bacterial endocarditis within 6 months (180 days) of procedure.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2011-03-09 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Leon, MD, Principal Investigator — Columbia University
Locations (53):
- United States (53):
  - Arkansas Heart Hospital/Clinic, Little Rock, Arkansas
  - Scripps Green Hospital, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Hospital, Denver, Colorado
  - Washington Hospital Center (WHC), Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida, Gainesville, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Indiana University Health-Methodist Hospital, Indianapolis, Indiana
  - The University of Iowa, Iowa City, Iowa
  - University of Louisville - Jewish Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City Mid America, Kansas City, Missouri
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Newark Beth Israel, Newark, New Jersey
  - North Shore University Hospital, NY, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Medical University of South Carolina Charleston, Charleston, North Carolina
  - East Carolina Heart Institute at East Carolina University, Greenville, North Carolina
  - The Christ Hospital, Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Austin Heart, PLLC, Austin, Texas
  - The Heart Hospital Baylor Plano, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - The University of Texas Health Science Center at Houston/Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio (UTHSCSA), San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shahim B, Redfors B, Lindman BR, Chen S, Dahlen T, Nazif T, Kapadia S, Gertz ZM, Crowley AC, Li D, Thourani VH, Kodali SK, Zajarias A, Babaliaros VC, Guyton RA, Elmariah S, Herrmann HC, Cohen DJ, Mack MJ, Smith CR, Leon MB, George I. Neutrophil-to-Lymphocyte Ratios in Patients Undergoing Aortic Valve Replacement: The PARTNER Trials and Registries. J Am Heart Assoc. 2022 Jun 7;11(11):e024091. doi: 10.1161/JAHA.121.024091. Epub 2022 Jun 3. PMID 35656983
- [Derived] Genereux P, Pibarot P, Redfors B, Bax JJ, Zhao Y, Makkar RR, Kapadia S, Thourani VH, Mack MJ, Nazif TM, Lindman BR, Babaliaros V, Vincent F, Russo M, McCabe JM, Gillam LD, Alu MC, Hahn RT, Webb JG, Leon MB, Cohen DJ. Evolution and Prognostic Impact of Cardiac Damage After Aortic Valve Replacement. J Am Coll Cardiol. 2022 Aug 23;80(8):783-800. doi: 10.1016/j.jacc.2022.05.006. Epub 2022 May 17. PMID 35595203
- [Derived] Chen S, Redfors B, O'Neill BP, Clavel MA, Pibarot P, Elmariah S, Nazif T, Crowley A, Ben-Yehuda O, Finn MT, Alu MC, Vahl TP, Kodali S, Leon MB, Lindman BR. Low and elevated B-type natriuretic peptide levels are associated with increased mortality in patients with preserved ejection fraction undergoing transcatheter aortic valve replacement: an analysis of the PARTNER II trial and registry. Eur Heart J. 2020 Feb 21;41(8):958-969. doi: 10.1093/eurheartj/ehz892. PMID 31883339
- [Derived] Summers MR, Leon MB, Smith CR, Kodali SK, Thourani VH, Herrmann HC, Makkar RR, Pibarot P, Webb JG, Leipsic J, Alu MC, Crowley A, Hahn RT, Kapadia SR, Tuzcu EM, Svensson L, Cremer PC, Jaber WA. Prosthetic Valve Endocarditis After TAVR and SAVR: Insights From the PARTNER Trials. Circulation. 2019 Dec 10;140(24):1984-1994. doi: 10.1161/CIRCULATIONAHA.119.041399. Epub 2019 Nov 6. PMID 31690104
- [Derived] Furer A, Chen S, Redfors B, Elmariah S, Pibarot P, Herrmann HC, Hahn RT, Kodali S, Thourani VH, Douglas PS, Alu MC, Fearon WF, Passeri J, Malaisrie SC, Crowley A, McAndrew T, Genereux P, Ben-Yehuda O, Leon MB, Burkhoff D. Effect of Baseline Left Ventricular Ejection Fraction on 2-Year Outcomes After Transcatheter Aortic Valve Replacement: Analysis of the PARTNER 2 Trials. Circ Heart Fail. 2019 Aug;12(8):e005809. doi: 10.1161/CIRCHEARTFAILURE.118.005809. Epub 2019 Aug 1. PMID 31525069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 53 sites in the US and Canada
Period: Overall Study
Arm/Group | TAVR - SAPIEN XT | TAVR - SAPIEN
Started | 284 | 276
As-Treated | 282 | 271
Valve-Implant | 280 | 263
Completed (One-year Follow-up) | 220 | 200
Not Completed | 64 | 76
Not completed — Death | 61 | 65
Not completed — Withdrawal by Subject | 3 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAVR - SAPIEN XT | TAVR - SAPIEN | Total
Number analyzed (Participants) | 284 | 276 | 560
Age, Continuous [Mean (Standard Deviation); unit: Years] | 84.0 (8.65) | 84.6 (8.61) | 84.3 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 134 | 277
  Male | 141 | 142 | 283
STS Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality and morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  units on a scale | 10.3 (5.38) | 11.0 (5.71) | 10.6 (5.55)
NYHA Class III/IV [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  Participants | 275 | 265 | 540
Coronary Artery Disease [Count of Participants; unit: Participants] | 186 | 186 | 372
Frailty [Count of Participants; unit: Participants] | 168 | 166 | 334

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Cause Mortality and/or Major Stroke and/or Rehospitalization
Description: All-Cause Mortality and/or Major Stroke and/or Rehospitalization at 1 Year
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | TAVR - SAPIEN XT | TAVR - SAPIEN
Number analyzed (Participants) | 284 | 276
participants | 105 | 102

2. Secondary Outcome: NYHA Classification - Change From Baseline
Description: New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
Time Frame: Baseline and 1 Year
Population: Please note that all the patients were not available for a NYHA functional assessment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TAVR - SAPIEN XT | TAVR - SAPIEN
Number analyzed (Participants) | 204 | 192
Units on a scale | -1.8 (0.92) | -1.7 (0.91)

3. Secondary Outcome: Total Aortic Regurgitation - Change From Baseline
Description: Total aortic regurgitation was assessed by the core lab as 'Grade 0' = None, 'Grade 1+' = Trace, 'Grade 2+' = Mild, 'Grade 3+' = Moderate, and 'Grade 4+' = Severe.
  Total regurgitation at one year was analyzed in the valve implant population.
Time Frame: 1 Year
Population: Please note that all the valve-implant population do not have echo data.
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | TAVR - SAPIEN XT | TAVR - SAPIEN
Number analyzed (Participants) | 172 | 155
Grade | 0.2 (1.38) | 0.1 (1.23)

4. Secondary Outcome: Effective Orifice Area - Change From Baseline
Time Frame: 1 Year
Population: Valve Implant Population; Please note that echo data was not available for all patients.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | TAVR - SAPIEN XT | TAVR - SAPIEN
Number analyzed (Participants) | 163 | 149
cm^2 | 0.9 (0.41) | 0.9 (0.38)

ADVERSE EVENTS:
Time Frame: Adverse event data are currently available and reported for all events at 1 year were reported at the time of database lock.
Description: All adverse events are site reported
  Only Valve-Implanted patients are reported for all adverse events (except for mortality).
Arm/Group | TAVR - SAPIEN XT | TAVR - SAPIEN
All-Cause Mortality (participants affected / at risk) | 10/282 | 12/271
Serious Adverse Events (participants affected / at risk) | 196/280 | 180/263
Other Adverse Events (participants affected / at risk) | 211/280 | 195/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR - SAPIEN XT (N=280) | TAVR - SAPIEN (N=263)
Abnormal lab value (Investigations) | 11 (13) | 7 (8)
Access site infection (Infections and infestations) | 5 (7) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 12 (13) | 14 (16)
Angina (Cardiac disorders) | 12 (14) | 0 (0)
Aortic root rupture (Vascular disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 33 (37) | 30 (31)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2) | 4 (5)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Cardiac arrest (Cardiac disorders) | 10 (10) | 17 (19)
Cardiac Tamponade/Pericardial Effusion (Cardiac disorders) | 4 (4) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 1 (1) | 0 (0)
Change in level of consciousness (Psychiatric disorders) | 2 (2) | 1 (1)
Cognitive Impairment (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3) | 5 (5)
Coronary Flow Obstruction/Transvalvular flow disturbance (General disorders) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Dementia (Psychiatric disorders) | 1 (1) | 0 (0)
Device Embolization (General disorders) | 1 (1) | 1 (1)
Device Migration (General disorders) | 3 (3) | 1 (1)
Dissection (Vascular disorders) | 10 (10) | 14 (14)
Distal embolization from vascular source (Vascular disorders) | 2 (2) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Edema (General disorders) | 1 (1) | 2 (2)
Embolization including air/calcific valve material or Thrombus (Vascular disorders) | 3 (3) | 4 (4)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Endocarditis (Cardiac disorders) | 2 (2) | 1 (1)
Exercise intolerance or weakness (General disorders) | 1 (1) | 1 (1)
Failure of percutaneous access site closure resulting in intervention (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 10 (11)
Fracture (Musculoskeletal and connective tissue disorders) | 9 (12) | 9 (10)
Gastro Intestinal Event (Gastrointestinal disorders) | 11 (11) | 10 (12)
Gastro Intestinal Event Nonhemorrhagic (Gastrointestinal disorders) | 6 (7) | 2 (2)
Genito Urinary Event (Renal and urinary disorders) | 4 (4) | 0 (0)
Genito Urinary Event Nonhemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Heart Failure / CHF / Low output Failure (Cardiac disorders) | 46 (64) | 39 (58)
Hematoma (Vascular disorders) | 5 (5) | 5 (5)
Hemiparesis (One sided body weakness) (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (One side limb weakness) (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 37 (41) | 30 (35)
Hemorrhagic Stroke (Nervous system disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 7 (7)
Ischemia (Vascular disorders) | 2 (2) | 0 (0)
Ischemic Stroke (Nervous system disorders) | 11 (11) | 8 (8)
Mitral Valve Injury or Insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Multi Organ Failure (General disorders) | 3 (3) | 1 (1)
Myocardial Infarction (Vascular disorders) | 6 (6) | 5 (5)
Non Structural Dysfunction (Cardiac disorders) | 6 (6) | 6 (6)
Other (General disorders) | 45 (56) | 42 (52)
Pain (General disorders) | 5 (5) | 7 (9)
Perforation (Vascular disorders) | 2 (2) | 9 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pseudoaneurysm (Vascular disorders) | 4 (4) | 8 (8)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (8)
Renal Insufficiency or Renal Failure (Renal and urinary disorders) | 16 (18) | 13 (16)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 15 (17)
Respiratory Infection (Infections and infestations) | 22 (25) | 17 (18)
Sepsis (Infections and infestations) | 14 (15) | 10 (11)
Stenosis (Cardiac disorders) | 2 (2) | 2 (2)
Structural Dysfunction (General disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 7 (7) | 8 (8)
TIA (Vascular disorders) | 1 (1) | 4 (4)
Thoracic aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Undetermined Stroke (Nervous system disorders) | 5 (5) | 2 (2)
Unknown cause of Death (General disorders) | 8 (8) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 12 (13) | 10 (11)
Ventricular rupture (Apical rupture) (Cardiac disorders) | 1 (1) | 0 (0)
Hemiplegia (One side limb weakness) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR - SAPIEN XT (N=280) | TAVR - SAPIEN (N=263)
Abnormal Lab Value (Investigations) | 49 (75) | 52 (77)
Anemia/Hemolytic Anemia (Blood and lymphatic system disorders) | 35 (45) | 36 (39)
Arrhythmia/Conduction System Injury (Defect) (Cardiac disorders) | 46 (52) | 41 (51)
Confusion (Psychiatric disorders) | 8 (8) | 16 (18)
Edema (Ear and labyrinth disorders) | 11 (11) | 18 (19)
Fall (Injury, poisoning and procedural complications) | 12 (14) | 19 (21)
Gastro Intestinal Event (Gastrointestinal disorders) | 19 (21) | 19 (22)
Hemorrhage (Vascular disorders) | 28 (33) | 30 (34)
Hypotension (Vascular disorders) | 12 (12) | 17 (17)
Non Structural Dysfunction (Injury, poisoning and procedural complications) | 13 (14) | 15 (16)
Pulmonary Effusion (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 18 (21)
Renal Insufficiency or Renal Failure (Renal and urinary disorders) | 22 (23) | 14 (16)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 14 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (17) | 18 (18)
Urinary Tract Infection (Renal and urinary disorders) | 28 (31) | 35 (45)
Other (General disorders) | 79 (105) | 87 (145)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other